CLINICAL TRIAL: NCT04586101
Title: iT-based Sports Therapy Application in Haemophilia
Acronym: iT-BaSTAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Dr. Thomas Hilberg (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. Dr. Thomas Hilberg, Chair holder - chair of sports medicine, University of Wuppertal
Organization: University of Wuppertal (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 35318939
Record Dates: First submitted 2020-07-28; First posted 2020-10-14 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Haemophilia; Sports Physical Therapy
Keywords: haemophilia; sports therapy; trainings application; home training
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training intervention (Experimental)
  Interventions: Device: Trainings application
- Control interverntion (No Intervention)

INTERVENTIONS:
Device: Trainings application — Participants have to train with the developed trainings application over six weeks. For this, individual training plans are implemented in the application based on orthopedic joint status and training recommendations of a sports scientist.
  Arms: Training intervention

SUMMARY:
Haemophilia is often associated with chronic pain, functional restrictions and negative consequences regarding the individual physical performance, especially on basic motoric skills, activities of daily life and quality of life. Caused by high benefits, physical activity is a fixed component and recommendation in the guidelines for the management of haemophilia. Several studies showed that goal-directed physical activity is feasible for patients with haemophilia (PwH) without any complications or bleeding episodes. Nevertheless, there are difficulties in the implementation of supervised sports therapy for PwH regarding local distributions and uncertainties concerning correct exercise execution on patients´ side and in the monitoring and adequate training regulation from long distances on the therapeutic side.

Aim of this project is a patient-related and participative development and pre-evaluation of a mobile application to generate an online-guided, individualized home training for PwH, followed by pre-evaluation in terms of a twelve weeks interventional phase. The intention of this project is to show, that a mobile device is an appropriate way to increase physical activity of PwH. Due to the development of an innovative trainings application, adapted to the needs of PwH, a larger number of patients should be reached and supported later on in participating on supervised physical exercise to improve the individual physical performance and therefore the quality of life. Additionally, with an individualized exercise program also adapted to the specific interests, needs and physical conditions, PwH at any age can be addressed. Furthermore, in cooperation with the patient, the medical staff will get systematic information of patients´ exercise activities to generate optimal factor and overall treatment patterns. In addition, on the basis of the mobile device PwH will be able to comprehend their individual exercise performance and to get an overview of the individual trainings progress and improvements of physical performance with the purpose to enhance the processes of self-motivation. Detailed instructions and information of exercise execution, need of exercise and physical adaptions to be achieved, will minimize complications and support patients´ self-confident for participating on exercise.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from moderate to severe haemophilia A or B
* submitted written consent to participate in the study
* approved sports capability and internet access

Exclusion Criteria:

* patients suffering from other bleeding disorders
* patients without written consent
* patients under 18 years of age
* patients without sports capability
* patients without internet access

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
frequency of physical activity | 12 weeks
  absolute number of completed physical activities
duration of physical activity | 12 weeks
  mean duration of completed physical activities

SECONDARY OUTCOMES:
score of subjective physical performance measured by the HEP-Test-Q | Day 1, 6 and 12 weeks
  questionnaire
score of subjective quality of life measured by the SF36 Health Survey | Day 1, 6 and 12 weeks
  questionnaire
pain intensity in score points measured by the German Pain Questionnaire | Day 1, 6 and 12 weeks
  questionnaire
health-related physical activity presented as metabolic equivalents of tasks | Day 1, 6 and 12 weeks
  questionnaire

OTHER OUTCOMES:
bleeding events | 12 weeks
  number
factor substitution in international units | 12 weeks
  administered international units of factor VIII or factor IX
frequency of factor substitution | 12 weeks
  absolute number of substitutions

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sports Medicine, University of Wuppertal, Wuppertal, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No